CLINICAL TRIAL: NCT04293965
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single-dose and Multiple-dose X842 in Healthy Subjects.
Brief Title: Single-dose and Multiple-dose X842 Phase 1 Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Sinorda Biomedicine Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: SND-X842-101; CTR20181666 (Other: Center for drug evaluation, NMPA)
Record Dates: First submitted 2020-02-07; First posted 2020-03-03 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers
Keywords: Potassium competitive acid blocker; Esophagitis; X842; Intragastric pH; Gastroesophageal reflux disease; GERD; Acid inhibition
MeSH Terms: conditions — Esophagitis; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: SAD, MAD and FE study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose Study (Experimental): Healthy subjects will be screened and different doses of X842 will be administered in a single dose to assess the safety, tolerability, PK and PD profile of X842.
  Interventions: Drug: Single ascending dose of X842
- Multiple Ascending Dose Study (Experimental): Healthy subjects will be screened and different doses of X842 will be administered in multiple doses to assess the safety, tolerability, PK and PD profile of X842. The dose ascending at this stage will be based on the results of the single dose tolerability study.
  Interventions: Drug: Multiple ascending dose of X842
- Food Effect Study (Experimental): A randomized, open label, single-dose, self-controlled, double-cycle, two-way crossover clinical trial.
  Interventions: Other: Food Effect

INTERVENTIONS:
Drug: Single ascending dose of X842 — A total of 7 dose groups will be set for the ascending dose: 5.6 mg, 12.5 mg, 25 mg, 50 mg, 100 mg, 150 mg, 225 mg. In the 5.6 mg dose group, 4 subjects will receive X842; in the 12.5 mg, 25 mg, 50 mg, 100 mg, 150 mg, 225 mg dose groups, 8 subjects in each group will receive X842. Each subject can only receive a certain dose level and cannot enter in multiple dose groups repeatedly.
  Other Names: X842
  Arms: Single Ascending Dose Study
Drug: Multiple ascending dose of X842 — Two dose groups will be set, including the groups receiving the recommended phase II dose and a higher dose; Eight subjects will be enrolled in each group, with half male and half female, who will receive X842 once daily for 5 consecutive days. Each subject can only receive a certain dose level and cannot enter in multiple dose groups repeatedly.
  Other Names: X842
  Arms: Multiple Ascending Dose Study
Other: Food Effect — Twelve subjects (appropriate ratio of male to female) screened for eligibility will be randomized into Group A and B. The 6 subjects in Group A will take the study drug (X842) in fasted condition and subject in Group B will take the study drug in fed condition in the 1st cycle. In the 2nd Cycle, subjects in Group A will take the study drug in fed condition, and subjects in Group B will take the study drug in fasted condition. The interval between the two cycles is at least 7 days.
  Other Names: X842
  Arms: Food Effect Study

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of X842 after administration of single and multiple doses in healthy subjects

DETAILED DESCRIPTION:
This is a single-center, open label, First-In-human (FIH), Phase I clinical study to evaluate the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) characteristics of single dose and multiple doses of X842 capsules in healthy subjects.

The study comprises a Single Ascending Dose (SAD) part, a Multiple Ascending Dose (MAD) part, and a Food Effect (FE) study.

ELIGIBILITY:
Inclusion Criteria:

1. Those aged 18-45 years old (inclusive the upper and lower limits).
2. Body weight of ≥ 50kg for male and ≥ 45kg for female , with a body mass index (BMI) of 19.0-26.0 kg/m2 (inclusive the upper and lower limits, BMI = weight (kg) / height (m) 2).
3. Understand and able to give written informed consent form for participation in this study voluntarily.

Those who fail to meet any of the above conditions shall not be enrolled.

Exclusion Criteria:

Those who meet any of the following conditions shall not be enrolled:

1. History of any clinically significant disease or disorder in cardiovascular system, respiratory system, digestive system, endocrine system, nervous/mental system, blood and lymphatic system, and musculoskeletal system according to the investigator.
2. Comprehensive physical examination, vital signs, laboratory test, 12-lead ECG, or chest X-ray examination (anteroposterior and lateral view) suggests that there are abnormalities that are determined by the investigator to be clinically significant.
3. Those who received helicobacter pylori eradication therapy within 6 months prior to the study drug administration;
4. The results of helicobacter pylori screening (C-14 urea breath test) is positive;
5. Any positive result for hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV), or Treponema pallidum antibody (TP-Ab).
6. History of any food or drug allergy, or any other history of allergic disease (such as asthma, urticaria, and eczematous dermatitis, etc.) considered as clinical significant by the investigator.
7. Subjects who had taken any drug within 2 weeks prior to screening, which may affect the results of the study according to the investigator.
8. History of drug abuse within 12 months prior to screening or positive urine drug result at screening.
9. Those who regularly drink alcohol within 6 months prior to screening, that is, more than 14 units of alcohol weekly (1 unit = 360 mL of beer or 45 mL of spirit with 40% alcohol or 150 mL of wine), or those who could not guarantee the abandonment of drinking during the study, or subjects with positive result of alcohol breath test.
10. Subjects who smoke more than 5 cigarettes daily within 3 months prior to screening or those could not guarantee the abandonment of smoking during the study.
11. Those who have participated in any other drug clinical trial within 3 months prior to screening (with the last visit date of the trial considered as the starting time for time counting).
12. Those who donated blood or blood products of ≥400ml or 2 units within 3 months or had lost of ≥400 mL blood within 6 months prior to screening.
13. Those who do not agree to stop alcohol drinking or caffeinated beverages within 48 hours before the study drug administration and throughout the whole trial, or do not agree to stop strenuous exercise or to avoid other factors that may affect the drug absorption, distribution, metabolism, or excretion.
14. Women who are pregnant or lactating, or who have a positive pregnancy test before the study drug administration; or those who could not or do not take the requested effective contraceptive measures accepted by the investigator during the trial.
15. Subjects with difficulties in venous blood collection, fear of needles or hemophobia.
16. Other conditions that may not be suitable for participating in the study judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Occurrence and frequency of AEs after single and multiple doses of X842. | Five Weeks
  Safety and tolerability will be assessed by occurrence and frequency of AEs. The adverse event assessment will follow the recommendations and grading system of Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Summary statistics will be applied.
Vital signs of body temperature | Five Weeks
Vital signs of blood pressure | Five Weeks
  Blood pressure measurements included systolic (mmHg) and diastolic (mmHg).
Vital signs of respiratory rate | Five Weeks
Physical Examination of height | Five Weeks
Physical Examination of weight | Five Weeks
Number of clinically significant changes in Electrocardiograms (ECGs) | Five Weeks
  The investigator or the sub-investigator interpreted the ECG using one of the following categories: "within normal limits", "abnormal but not clinically significant", or "abnormal and clinically significant".
Number of Clinically significant changes in lab assessment of blood serum | Five Weeks
Number of Clinically significant changes in the lab assessment of blood | Five Weeks
Number of Clinically significant changes in the lab assessment of urine | Five Weeks

SECONDARY OUTCOMES:
Measurement of the PK profile (Cmax) | Up to 48 hours after dosing
  To assess the Maximum Plasma Concentration (Cmax)
Measurement of the PK profile (t1/2) | Up to 48 hours after dosing
  To assess the plasma half life (t1/2) of drug
Measurement of the PD profile (intragastric pH) | Up to 24 hours after dosing
  To assess and characterize the PD profile with measurements of intragastric pH

CONTACTS AND LOCATIONS:
Overall Officials: Pingsheng Hu, Ph.D, Study Chair — Jiangsu Sinorda Biomedicine Co., Ltd
Locations (1):
- The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Serag HB, Sweet S, Winchester CC, Dent J. Update on the epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2014 Jun;63(6):871-80. doi: 10.1136/gutjnl-2012-304269. Epub 2013 Jul 13. PMID 23853213
- [Background] Yuan Y, Hunt RH. Evolving issues in the management of reflux disease? Curr Opin Gastroenterol. 2009 Jul;25(4):342-51. doi: 10.1097/MOG.0b013e32832c1504. PMID 19417644
- [Background] Dent J, Kahrilas PJ, Hatlebakk J, Vakil N, Denison H, Franzen S, Lundborg P. A randomized, comparative trial of a potassium-competitive acid blocker (AZD0865) and esomeprazole for the treatment of patients with nonerosive reflux disease. Am J Gastroenterol. 2008 Jan;103(1):20-6. doi: 10.1111/j.1572-0241.2007.01544.x. PMID 18184117
- [Background] Kahrilas PJ, Dent J, Lauritsen K, Malfertheiner P, Denison H, Franzen S, Hasselgren G. A randomized, comparative study of three doses of AZD0865 and esomeprazole for healing of reflux esophagitis. Clin Gastroenterol Hepatol. 2007 Dec;5(12):1385-91. doi: 10.1016/j.cgh.2007.08.014. Epub 2007 Oct 22. PMID 17950677
- [Background] Nilsson, Albrektson E, Rydholm H, Rohss K, Alin MH, Hasselgren G. Tolerability, Pharmacokinetics and Effects on Gastric Acid Secretion After Single Oral Doses of the Potassium-Competitive Acid Blocker (P-CAB) AZD0865 in Healthy Male Subjects. Gastroenterology 2005 Volume 128, Issue 4, Supplement 2.